CLINICAL TRIAL: NCT02609685
Title: Active Surveillance of Papillary Thyroid Microcarcinoma
Acronym: PMCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Allen Ho, Director, Head and Neck Cancer Program and Co-Director, Thyroid Cancer Program, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIT2014-13-Ho-PMCAS
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Papillary Thyroid Microcarcinoma
Keywords: Thyroid cancer; Active surveillance; PTMC
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma; Thyroid Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Surveillance (Other): Active surveillance instead of standard of care immediate surgery. Patients will be closely monitored every six months until disease is stable for a two-year period and then annually thereafter.
  Interventions: Other: Active Surveillance
- Immediate Surgery (No Intervention): Patients who choose to get surgery immediately after diagnosis may choose to enroll in a questionnaire sub-study that will compare quality of life and anxiety scores to patients who enroll in the active surveillance study. This is considered "no intervention" because the protocol is not directing treatment. Surgery is the standard treatment for papillary thyroid microcarcinoma.

INTERVENTIONS:
Other: Active Surveillance — Subjects will be actively observed for disease progression (condition worsens) instead of receiving immediate surgery, considered standard of care.
  Arms: Active Surveillance

SUMMARY:
The purpose of this study is to better understand the outcomes of active surveillance (observation) instead of immediate surgery, which is the current standard of care for papillary thyroid microcarcinoma (PTMC). Patients with a 1.5 cm or smaller thyroid nodule(s) with papillary thyroid carcinoma will be eligible for the study.

DETAILED DESCRIPTION:
The incidence of thyroid cancer has more than doubled in the last 30 years in the United States, Europe, Canada, and South America. Since nearly 50% of this increase is attributable to papillary thyroid microcarcinomas (PTMC), it appears that greater detection and diagnosis of previously subclinical disease is a major factor driving this dramatic rise.

The primary objective is to estimate the rate of disease progression (growth of primary tumor or development of loco-regional/distant metastases) over a 3, 5, and 10-year period in a series of PTMC patients followed with active surveillance in the United States.

Patients who opt for immediate surgery can participate in a sub-study looking at quality of life and anxiety measures as compared to those patients who enroll in the active surveillance main study. Patients who enroll in active surveillance can choose to have surgery at any time that they and their treating physician feel that it is in their best interest.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Bethesda V or VI thyroid nodules with papillary thyroid carcinoma or high clinical suspicion, or pathologically confirmed Bethesda III or IV nodules with BRAF mutation.
* 2.0 cm or smaller nodules by ultrasonographic criteria
* Ability to understand and the willingness to sign a written informed consent and HIPAA Authorization form
* Must be able to read and write English fluently to participate in the questionnaire portion of the study

Exclusion Criteria:

* High-grade or poorly differentiated PTC variants
* Central or lateral neck lymphadenopathy suspicious for PTC
* Unfavorable nodule location (e.g. Near dorsal surface (by recurrent laryngeal nerve); Adjacent to trachea (risk of cartilage invasion)
* History of radiation to neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2016-05-13 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of disease progression | From time of diagnosis up to10 years of follow-up

SECONDARY OUTCOMES:
Percentage of subjects that will elect surgery despite absence of clinical progression | From time of diagnosis up to 10 years of follow-up
Impact of TSH suppression on thyroid nodule growth (in cm) as measured by ultrasound | Five years
Identify the clinicopathologic features associated with disease progression in papillary thyroid microcarcinoma patients followed with active surveillance | Five years
Identify the genetic factors associated with an increased risk of disease progression | Five years
  At any time subjects who have enrolled in the active surveillance study can opt to have surgery. Data will be taken from diagnosis to just after surgery.
Quality of life score as measured by City of Hope Quality of Life Scale | Up to five years
Anxiety score as measured by Memorial Anxiety Scale | Up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Allen Ho, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho AS, Kim S, Zalt C, Melany ML, Chen IE, Vasquez J, Mallen-St Clair J, Chen MM, Vasquez M, Fan X, van Deen WK, Haile RW, Daskivich TJ, Zumsteg ZS, Braunstein GD, Sacks WL. Expanded Parameters in Active Surveillance for Low-risk Papillary Thyroid Carcinoma: A Nonrandomized Controlled Trial. JAMA Oncol. 2022 Sep 15;8(11):1588-96. doi: 10.1001/jamaoncol.2022.3875. Online ahead of print. PMID 36107411